CLINICAL TRIAL: NCT06520787
Title: DAta-driven personaLIzation of a digitAl Health Solution to Support Family Caregivers of Children With Chronic Conditions
Acronym: DALIA
Status: Recruiting | Type: Observational
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Hospital Universitario Miguel Servet, Zaragoza (Unknown); University of Valencia (Other); University of Seville (Other)
Responsible Party: Sponsor
Other Study IDs: DAL-CLI-24-001
Record Dates: First submitted 2024-07-04; First posted 2024-07-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Childhood
Keywords: Obesity; Digital health; Treatment satisfaction; pharmacological treatment for obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — 2-amino-3-cyano-6-methyl-5-(3,4-dimethoxyphenyl)pyridine; Drug Therapy; Adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: 40 families with children already receiving pharmacological therapy as per clinical indication will be asked to use the ACDP® for obesity. We will track their progress with the digital intervention for ten months, and there will be a 2-month follow-up (total 12 months)
  Interventions: Combination Product: ACDP® and pharmacological treatment for obesity

INTERVENTIONS:
Combination Product: ACDP® and pharmacological treatment for obesity — 40 Families of children with obesity that are already undergoing treatment and are willing to join a combined intervention. After the recruitment, the family will join Adhera Caring Digital Program® for 10 months. The combined intervention (digital and pharmacological intervention) will last one year, and there will be a 2-month follow-up. During the whole study (12 months, from recruiting to the end of follow-up) participants will wear a smartwatch (Fitbit or similar).

SUMMARY:
The goal of this feasibility study is to explore the needs of families with children with obesity and evaluate the impact of a combined intervention (children with obesity receiving pharmacological therapy in combination with the Adhera Caring Digital Program®) on treatment satisfaction, adherence, and mood. The main objectives are:

* To evaluate the impact of the treatment combination (ACDP® and pharmacological treatment) in terms of satisfaction, engagement, adherence and mood, in families with children with obesity.
* To better understand the educational and support needs of the families of children with obesity while under treatment and lifestyle changes.

Participants will:

* Use the Adhera Caring Digital Program® (ACDP®) for obesity, which includes digital therapeutic software, personalized messages, and educational materials.
* Take pharmacological treatment as prescribed for one year.
* Wear activity wristbands/watches to collect biometric data.
* Attend monthly clinic visits for assessments and monitoring.
* Complete psychometric questionnaires to measure satisfaction, adherence, and emotional outcomes.
* Engage in chat-based communication and video conferencing with health coaches for support and monitoring.

ELIGIBILITY:
Inclusion criteria:

* Caregivers of children between 13 and 18 years who are diagnosed with obesity and undergoing treatment according to the approved label by AEMPS1 (adolescents with obesity aged 12 years and older with an initial BMI at the 95th percentile or greater for age and sex).
* Families of children with obesity who have been under pharmacological treatment before screening. This includes treatment with any of the following medications orlistat, metformin, liraglutide, semaglutide.
* Participants who are willing to join ACDP® for 10 months and can interact with a smartphone during that time.
* The family is willing to complement the pharmacological obesity treatment with a digital intervention.
* Participants (patients and their caregivers) must be willing to use wearables for the entire length of the study.
* Parents previously using a wearable will agree not to use it during the length of the study, as their wearable account must be synched to the patient's device. Further, they may need to agree on changing the account data for height, weight, and gender in their Google account.

Exclusion criteria:

* Families not fluent in Spanish.
* Families of children with obesity and comorbidities.
* Families of children with secondary causes of obesity (i.e., hypothalamic, genetic or endocrine causes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of the study (caregivers) will be recruited from the Pediatric Endocrinology unit at the Miguel Servet Children's University Hospital. This public hospital provides pediatric health attention to the regional area of Zaragoza (Spain), which covers a total of 367.110 inhabitants.
  Families of children with obesity that are already undergoing treatment and are willing to join a combined intervention.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction | Day 1 to Day 365
  Treatment satisfaction measured by Treatment Expectation Scale/Treatment Satisfacyion Scale. Minimum Value: 0. Maximum Value: 10. Interpretation: Higher scores indicate better outcomes (greater treatment expectation/satisfaction).
Treatment adherence 1 | Day 1 to Day 365
  Treatment adherence measured by injection (self-reported). Unit of measure: Number of injections (quantitative data)
Treatment adherence 2 | Day 1 to Day 365
  Treatment adherence measured by changes in nutritional compliance (self-reported). Unit of measure: Description of diet (qualitative data).
Treatment adherence 3 | Day 150 to Day 365
  Treatment adherence measured by discontinuation (and reasons behind it). Unit of measure: Incidence of discontinuation with categorized reasons.

SECONDARY OUTCOMES:
Emotional outcome 1 | Baseline (Day 1) to Day 365
  These tend to be sensitive to change in short-term and will include distress assessed by the Depression Anxiety and Stress Scale (DASS-21) and the distress thermometer. Minimum Value: 0. Maximum Value: 63. Interpretation: Higher scores indicate worse outcomes (greater levels of depression, anxiety, and stress).
Emotional outcome 2 | Baseline (Day 1) to Day 365
  These tend to be sensitive to change in short-term and will include Weight Self-Stigma Questionnaire (S-WSSQ). Minimum Value: 12. Maximum Value: 60. Interpretation: Higher scores indicate worse outcomes (greater self-stigma related to weight).
Emotional outcome 3 | Baseline (Day 1) to Day 365
  These tend to be sensitive to change in short-term and will include perceived self-efficacy assessment by the General Self-Efficacy Scale (GSE). Minimum Value: 10. Maximum Value: 40. Interpretation: Higher scores indicate better outcomes (greater self-efficacy).
Health-related Quality of Life (HrQoL) | Baseline (Day 1) to Day 365
  Quality of life tends to change over longer periods of time, and often do require follow-ups of 6 months or one year. However, some dimensions (e.g. mental) are estimated to change faster in shorter periods. HrQoL will be assessed with regard to the children by the caregivers' perspective from the KIDSCREEN-10. Minimum Value: 10. Maximum Value: 50. Interpretation: Higher scores indicate better outcomes (better health-related quality of life).
Levels of physical activity | Baseline (Day 1) to Day 365
  Life-style questionnaires on Levels of physical activity (APALQ; Assessment of Physical Activity Levels Questionnaire ). Minimum Value: Varies based on questionnaire design. Maximum Value: Varies based on questionnaire design. Interpretation: Higher scores generally indicate better outcomes (higher levels of physical activity).
Height | Baseline (Day 1) to Day 365
  From bioimpedance scale. Standard medical measurement. Unit of measure: meters.
Weight | Baseline (Day 1) to Day 365
  From bioimpedance scale. Standard medical measurement. Unit of measure: kilograms.
Body Mass Index (BMI) | Baseline (Day 1) to Day 365
  From bioimpedance scale. Calculated from height and weight. Unit of measure: kg/m²
Blood pressure | Baseline (Day 1) to Day 365
  Standard pressure measurement. Unit of measure: mmHg.
Time since diagnosis | Baseline (Day 1) to Day 365
  From patient medical records or self-reported data. Unit of measure: weeks, months or years.
Previous obesity treatments | Baseline (Day 1) to Day 365
  From patient medical records and self-reported data. Unit of measure: Description of treatment (qualitative data).
Cholesterol levels | Baseline (Day 1) to Day 365
  Blood test results. Unit of measure: mg/dL
Complications | Baseline (Day 1) to Day 365
  From patient medical records or self-reported. Unit of measure: Incidence and type of complications (qualitative data)
Step count | Baseline (Day 1) to Day 396
  From wearable device. Unit of measure: number of steps per day.
Physical activity levels | Baseline (Day 1) to Day 300
  From wearable device. Unit of measure: minutes of moderate to vigorous activity per day.
Sleep quality | Baseline (Day 1) to Day 300
  From wearable device. Unit of measure: Sleep score or duration and quality of sleep (hours and sleep stages).
Heart rate | Baseline (Day 1) to Day 300
  From wearable device. Unit of measure: average resting heart rate (beats per minute).
6-minute walk test performance | Baseline (Day 1) to Day 365
  Standardized 6-minute walk test. Unit of measure: distance covered in meters.
System Usability | Day 150 to 300
  Measures the perceived usability of ACDP. Minimum Value: 0. Maximum Value: 10. Interpretation: Higher scores indicate better perceibed usability

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No